CLINICAL TRIAL: NCT00977327
Title: Comparison of Two Neuro-navigational Systems for Resection-control of Intra-axial Brain Tumors. The PoleStarN-20 Intra-operative Magnet Resonance Imager and the Mison SonoWand Intra-operative Ultrasound System
Brief Title: Comparison of Neuro-navigational Systems for Resection-Control of Brain Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Andrew Kanner MD, Department of Neurosurgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-09-AK-0351
Record Dates: First submitted 2009-08-30; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Glioma
Keywords: Glioma; Intraoperative MR; Intraoperative Ultrasound; resection; Intraoperative navigation; Extent of resection
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraoperative MR (Other): Use of intraoperative MR during resection of intraaxial tumor, Glioma
  Interventions: Device: Intraoperative MR (PoleStar N-20, Medtronics)
- Intraoperative Ultrasound (Other): Use of intraoperative ultrasound during resection of intraaxial tumor, Glioma
  Interventions: Device: Intraoperative Ultrasound (Sonowand, Mison)

INTERVENTIONS:
Device: Intraoperative MR (PoleStar N-20, Medtronics) — intraoperative imaging for resection control of intraaxial brain lesions
  Other Names: PoleStar N-20, Medtronics
  Arms: Intraoperative MR
Device: Intraoperative Ultrasound (Sonowand, Mison) — intraoperative imaging for resection control of intraaxial brain lesions
  Other Names: Sonowand, Mison
  Arms: Intraoperative Ultrasound

SUMMARY:
Purpose:

* Improvement of extent of resection by the use of intraoperatively acquired image data sets to navigate.
* Better define the role of different intra-operative imaging modalities, used to update the navigational data set, in aiding the surgeon during resection of intra-axial brain lesions.
* To examine the cost-effectiveness of different intraoperative navigational systems as a function of operative time and Operative time (Surgery including imaging)

There is increasing neuro-oncological evidence that extent of resection might have an impact in particular in low-grade lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have neuro-radiological evidence of a brain lesion. Eligible are all histological types of brain lesions.
* > 18 years of age.
* Male and female.
* Patient must be a surgical candidate, according to general anesthetic and neurosurgical criteria.
* Patient should be able to undergo MRI.
* Informed consent as per protocol.

Exclusion Criteria:

* Patient unwilling to undergo surgery for resection of brain tumor.
* Patient medically not eligible to undergo craniotomy. (Medical contraindication).
* Patient has a medical contraindication or is unwilling to undergo MRI scanning (pacemaker, other metal device ot parts in head or body,).
* Kidney function compromise (Creatinine values > 1.4 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The primary end point of the study is assessment and comparison of intra-operative Magnet Resonance Imaging and ultrasound to better define its impact on the extent of resection. | 72 hours

SECONDARY OUTCOMES:
Secondary end points should identify criteria for selecting the right system for a specific patient (Patient selection), and cost-effectiveness. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kanner, MD, Principal Investigator — Tel-Aviv Sorasky Medical Center
Locations (1):
- Tel-Aviv Sorasky MC, Tel Aviv, Israel